CLINICAL TRIAL: NCT01504386
Title: Effekt of Transversus Abdominis Plane (TAP) Block After Robot-assisted Laparocopic Hysterectomy
Brief Title: Transversus Abdominis Plane Block After Robot-assisted Laparocopic Hysterectomy
Acronym: TAP-block
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Due to local restructering, further recruting was not possible
Sponsor: Copenhagen University Hospital at Herlev (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SM1-HT-2011
Record Dates: First submitted 2011-12-30; First posted 2012-01-05 (Estimated); Last update posted 2013-08-22 (Estimated); Status verified 2013-08

CONDITIONS: Hysterectomy
MeSH Terms: interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TAP block (Experimental): TAP block with ropivacaine
  Interventions: Procedure: TAP block
- Placebo TAP block (Placebo Comparator): Sham block with saline
  Interventions: Procedure: Placebo TAP block

INTERVENTIONS:
Procedure: TAP block — Bilateral UL-guided TAP block with 20 ml of ropivacaine 0.5 %
  Other Names: Naropin 0.5%
  Arms: TAP block
Procedure: Placebo TAP block — Bilateral placement of 20 ml of saline 0.9 % in the transversus abdominis plane
  Other Names: Saline 0.9%
  Arms: Placebo TAP block

SUMMARY:
The purpose of this study is to investigate the effectiveness of Transversus Abdominis Plane (TAP) block as a part of a multimodal postoperative pain management after robot-assisted laparoscopic hysterecomy.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80
* BMI 17-40
* Written consent
* Can cooperate

Exclusion Criteria:

* Drug and alcohol abuse
* Consumption of opioids
* Drug allergy
* Infection at insertion point of needle

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2011-12; Primary Completion 2013-03 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Total opioid consumption | 0-24 hours
  Opioid consumption via PCA-pump

SECONDARY OUTCOMES:
Pain during rest and cough | 1,2,4,8,18 and 24 hours
  VAS-pain score at rest and at cough
Postoperative nausea and vomiting | 1,2,4,8,18 and 24 hours
  Nausea score 0-3 No. of vomits

CONTACTS AND LOCATIONS:
Overall Officials: Henrik Torup, MD, Principal Investigator — Herlev University Hospital, Copenhagen
Locations (1):
- Herlev Univerity Hospital, Department of Anaesthesia, Herlev, Denmark